CLINICAL TRIAL: NCT02203955
Title: Prevention of Pouchitis With Short-Chain Fructooligosaccharide Therapy, A Double-Blind, Placebo-Controlled Trial
Brief Title: Study of Sc-FOS for Pouchitis Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Laura E. Raffals, M.D, Assistant Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14-001220
Record Dates: First submitted 2014-07-16; First posted 2014-07-30 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Pouchitis
MeSH Terms: conditions — Pouchitis | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short-Chain Fructooligosaccharide (Active Comparator): 4 chews (8.0 g scFOS) orally per day for 12 months
  Interventions: Drug: Short-Chain Fructooligosaccharide
- Maltodextrin (Placebo Comparator): 4 chews (maltodextrin) daily for 12 months
  Interventions: Drug: Maltodextrin

INTERVENTIONS:
Drug: Short-Chain Fructooligosaccharide — 4 chews (8.0 g scFOS) orally for 12 months
  Arms: Short-Chain Fructooligosaccharide
Drug: Maltodextrin — 4 chews (maltodextrin) daily for 12 months
  Arms: Maltodextrin

SUMMARY:
The main objective is to compare prebiotic therapy with placebo for the prevention of pouchitis after closure of diverting ileostomy in patients with an ileal pouch anal anastomosis. This study will also characterize the effects of prebiotics on the fecal microbiota and fecal microbial metabolites and correlate these effects with the primary outcome of development of pouchitis.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-65 years.
2. History of ulcerative colitis
3. Ileostomy closure after IPAA
4. Ability to give appropriate consent

Exclusion Criteria:

1. Crohn's disease.
2. Perianal disease (including abscess, fissure, or stricture)
3. Pregnancy
4. Lactation
5. Concurrent treatment for IBD or pouchitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Mean Change in Pouchitis Disease Activity Index (PDAI) at One Year | baseline, 1 year
  In the PDAI, an overall score is calculated from three separate six-point scales comprising of clinical symptoms, endoscopic findings and histological changes. The PDAI incorporates histological features of acute inflammation, and establishes a cut-off of seven for differentiation between 'pouchitis (≥7 points) and 'no pouchitis' (<7 points).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Raffals, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials